CLINICAL TRIAL: NCT01728623
Title: A Phase 2 Study of E7080 in Subjects With Advanced Thyroid Cancer
Brief Title: A Study of E7080 in Subjects With Advanced Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-J081-208
Record Dates: First submitted 2012-09-07; First posted 2012-11-20 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-07

CONDITIONS: Thyroid Cancer
Keywords: Thyroid cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — lenvatinib

ARMS (1):
- E7080 (Experimental)
  Interventions: Drug: E7080 capsule

INTERVENTIONS:
Drug: E7080 capsule — E7080 is administered as continuous once daily dosing in an uncontrolled manner

SUMMARY:
This study is to evaluate the safety, efficacy, and pharmacokinetics of E7080 when orally administered once daily (QD) in subjects with advanced thyroid cancer.

ELIGIBILITY:
Inclusion criteria

1. Histologically or clinically diagnosed with thyroid cancer
2. Eastern Cooperative Oncology Group Performance Status (ECOG-PS) 0-2
3. Adequate laboratory values/organ function tests

Exclusion criteria

Participants with following complication or disease history

1. Brain metastasis
2. Systemic severe infection
3. Significant cardiovascular impairment
4. QTc greater than 480 milliseconds
5. Active hemoptysis
6. Bleeding or thrombotic disorders
7. Having greater than 1+ proteinuria on urine dipstick testing will undergo 24 hour urine collection for quantitative assessment of proteinuria
8. Gastrointestinal malabsorption or any other condition in the opinion of the investigator that might affect the absorption of E7080
9. Major surgery within 3 weeks before enrollment
10. With co-existing effusion requiring drainage

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-09-03 (Actual); Primary Completion 2015-07-09 (Actual); Study Completion 2015-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Kashiwa, Chiba
  - Kobe, Hyōgo
  - Koto-ward, Tokyo

REFERENCES:
- [Derived] Takahashi S, Kiyota N, Yamazaki T, Chayahara N, Nakano K, Inagaki L, Toda K, Enokida T, Minami H, Imamura Y, Fukuda N, Sasaki T, Suzuki T, Ikezawa H, Dutcus CE, Tahara M. A Phase II study of the safety and efficacy of lenvatinib in patients with advanced thyroid cancer. Future Oncol. 2019 Mar;15(7):717-726. doi: 10.2217/fon-2018-0557. Epub 2019 Jan 14. PMID 30638399
- [Derived] Tahara M, Kiyota N, Yamazaki T, Chayahara N, Nakano K, Inagaki L, Toda K, Enokida T, Minami H, Imamura Y, Sasaki T, Suzuki T, Fujino K, Dutcus CE, Takahashi S. Lenvatinib for Anaplastic Thyroid Cancer. Front Oncol. 2017 Mar 1;7:25. doi: 10.3389/fonc.2017.00025. eCollection 2017. PMID 28299283

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 4: Lenvatinib (MTC, DTC, ATC): Participants received 24 milligram (mg) lenvatinib capsule (two 10 mg capsules and one 4 mg capsule) orally once daily in the morning in a 28-day treatment cycle for until participant met one or more discontinuation criteria by individual participant. Arm 4 included all treated participants (differentiated thyroid cancer [DTC], medullary thyroid cancer [MTC], and anaplastic thyroid cancer [ATC]).
Period: Overall Study
Arm/Group | Arm 4: Lenvatinib (MTC, DTC, ATC)
Started | 51
DTC | 25
MTC | 9
ATC | 17
Completed | 23
Not Completed | 28
Not completed — Disease progression | 26
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least one dose of study drug and had at least one postbaseline safety evaluation.
Groups:
- Lenvatinib (Arm 1): Participants received 24 mg lenvatinib capsule (two 10 mg capsules and one 4 mg capsule) orally once daily in the morning in a 28-day treatment cycle for until participant met one or more discontinuation criteria by individual participant. Arm 1 included participants with DTC.
- Lenvatinib (Arm 2): Participants received 24 mg lenvatinib capsule (two 10 mg capsules and one 4 mg capsule) orally once daily in the morning in a 28-day treatment cycle for until participant met one or more discontinuation criteria by individual participant. Arm 2 included participants with MTC.
- Lenvatinib (Arm 3): Participants received 24 mg lenvatinib capsule (two 10 mg capsules and one 4 mg capsule) orally once daily in the morning in a 28-day treatment cycle for until participant met one or more discontinuation criteria by individual participant. Arm 3 included participants with ATC.
- Total: Total of all reporting groups
Arm/Group | Lenvatinib (Arm 1) | Lenvatinib (Arm 2) | Lenvatinib (Arm 3) | Total
Number analyzed (Participants) | 25 | 9 | 17 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (12.34) | 60.6 (13.70) | 63.4 (11.40) | 59.8 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 3 | 11 | 30
  Male | 9 | 6 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Only TEAEs are included in the summary. For detailed list of adverse events (AEs), see the AE section. For each participant, only one TEAE in the same category was counted and for multiple TEAEs with different Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v 4.0) grades, only the event with the highest grade was reported. All AEs were graded using CTCAE v 4.0, except for alopecia and infertility.
Time Frame: Screening visit to 30 days after the last dose of study drug, or assessed up to 3 years
Population: Safety population included all participants who received at least one dose of study drug and had at least one postbaseline safety evaluation.
Measure: Number; unit: Percentage of participants
Groups:
- Arm 4: Lenvatinib (DTC, MTC, ATC): Participants received 24 mg lenvatinib capsule (two 10 mg capsules and one 4 mg capsule) orally once daily in the morning in a 28-day treatment cycle for until participant met one or more discontinuation criteria by individual participant. Arm 4 included all treated participants (DTC, MTC and ATC).
Arm/Group | Arm 4: Lenvatinib (DTC, MTC, ATC)
Number analyzed (Participants) | 51
Percentage of participants
  TEAEs | 100.0
  CTCAE Grade 3 or 4 TEAEs | 82.4
  Serious TEAEs | 52.9
  TEAEs leading to study drug withdrawal | 2.0
  TEAEs leading to study drug reduction | 96.1
  TEAEs leading to study drug interruption | 66.7

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from (1) the date of randomization to the date of first documentation of disease progression based on Investigator and Independent Review Committee assessments according to Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST v1.1), or (2) death, whichever came first. Disease progression for the MTC group was measured using computed tomography (CT) or magnetic resonance imaging (MRI) on targeted tumors. Disease progression per RECIST v1.1 was defined as at least a 20 percent (%) relative increase and 5 millimeter (mm) absolute increase in the sum of diameters of target lesions (taking as reference the smallest sum on study), recorded since the treatment started or the appearance of 1 or more new lesions. Summarized by the Kaplan-Meier method using median time with 95% confidence interval (CI).
Time Frame: From first date of study treatment until progression of disease or date of death from any cause, whichever comes first, assessed up to 34 months
Population: Full analysis set included all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib (Arm 1) | Lenvatinib (Arm 2) | Lenvatinib (Arm 3)
Number analyzed (Participants) | 25 | 9 | 17
Months | 25.8 [18.4 to NA] — Upper limit of 95% confidence interval (CI) could not be calculated since insufficient number of participants had an event. | 9.2 [1.8 to NA] — Upper limit of 95% confidence interval (CI) could not be calculated since insufficient number of participants had an event. | 7.4 [1.7 to 12.9]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose of study treatment to the date of death from any cause. If death was not observed for a participant, the survival time was censored at the date the participant was last known alive or the data cutoff date (whichever occurred first). Summarized by the Kaplan-Meier method using median time with 95% CI.
Time Frame: From study start until date of death from any cause, assessed up to 34 months
Population: Full analysis set included all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib (Arm 1) | Lenvatinib (Arm 2) | Lenvatinib (Arm 3)
Number analyzed (Participants) | 25 | 9 | 17
Months | 31.8 [31.8 to NA] — Upper limit of 95% CI could not be calculated since insufficient number of participants had an event. | 12.1 [3.8 to NA] — Upper limit of 95% CI could not be calculated since insufficient number of participants had an event. | 10.6 [3.8 to 19.8]

4. Secondary Outcome: Best Overall Response (BOR)
Description: BOR was defined as the best response observed between the time of first dose and the study completion, assessed by either of complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), or not evaluable (NE). Tumor assessment was performed by the investigator using RECIST 1.1. The CR and PR were determined only when these responses met each criterion even after 28 days from the time observed. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had to have reduction in short axis to less than 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as greater than or equal to 7 weeks for DTC and MTC, greater than or equal to 3 weeks for ATC.
Time Frame: Date of first dose of study treatment to CR, PR, SD, PD, or NE, assessed up to 34 months
Population: Full analysis set included all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Lenvatinib (Arm 1) | Lenvatinib (Arm 2) | Lenvatinib (Arm 3)
Number analyzed (Participants) | 25 | 9 | 17
Percentage of participants
  CR | 0 | 0 | 0
  PR | 68.0 | 22.2 | 23.5
  SD | 32.0 | 77.8 | 70.6
  PD | 0 | 0 | 5.9
  NE | 0 | 0 | 0

5. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who had BOR of CR or PR. Tumor assessment was performed by the investigator using RECIST 1.1. ORR based on the investigator assessment was provided with a corresponding exact 95% CI which was calculated using exact method of binomial distribution.
Time Frame: Date of CR or PR to date of PD or death (whichever was first), assessed up to 34 months
Population: Full analysis set included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenvatinib (Arm 1) | Lenvatinib (Arm 2) | Lenvatinib (Arm 3)
Number analyzed (Participants) | 25 | 9 | 17
Percentage of participants | 68.0 [46.5 to 85.1] | 22.2 [2.8 to 60.0] | 23.5 [6.8 to 49.9]

6. Secondary Outcome: Disease Control Rate (DCR)
Description: The DCR was defined as the percentage of participants who had BOR of CR, PR, or SD. Tumor assessment was performed by the investigator using RECIST 1.1. DCR based on the investigator assessment was provided with a corresponding exact 95% CI which was calculated using exact method of binomial distribution.
Time Frame: Date of CR, PR, or SD to date of PD or death (whichever was first), assessed up to 34 months
Population: Full analysis set included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenvatinib (Arm 1) | Lenvatinib (Arm 2) | Lenvatinib (Arm 3)
Number analyzed (Participants) | 25 | 9 | 17
Percentage of participants | 100.0 [86.3 to 100.0] | 100.0 [66.4 to 100.0] | 94.1 [71.3 to 99.9]

7. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: The CBR was defined as the percentage of participants who had BOR of CR, PR, or durable SD (dSD). Tumor assessment was performed by the investigator using RECIST 1.1. Durable stable disease was defined as SD lasting greater than or equal to 23 weeks for DTC and MTC, greater than or equal to 11 weeks for ATC. A 95% CI was calculated using exact method of binomial distribution.
Time Frame: Date of CR, PR, or dSD to date of PD or death (whichever was first), assessed up to 34 months
Population: Full analysis set included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenvatinib (Arm 1) | Lenvatinib (Arm 2) | Lenvatinib (Arm 3)
Number analyzed (Participants) | 25 | 9 | 17
Percentage of participants | 84.0 [63.9 to 95.5] | 77.8 [40.0 to 97.2] | 70.6 [44.0 to 89.7]

ADVERSE EVENTS:
Time Frame: AEs were collected for up to 3 years
Description: Safety population included all participants who received at least one dose of study drug and had at least one postbaseline safety evaluation.
Arm/Group | Arm 4: Lenvatinib (DTC, MTC, ATC)
All-Cause Mortality (participants affected / at risk) | 4/51
Serious Adverse Events (participants affected / at risk) | 27/51
Other Adverse Events (participants affected / at risk) | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 4: Lenvatinib (DTC, MTC, ATC) (N=51)
Diarrhoea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 1
Oedema peripheral (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Respiratory tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 7
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vagus nerve disorder (Nervous system disorders) | 1
Vocal cord paralysis (Nervous system disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 4: Lenvatinib (DTC, MTC, ATC) (N=51)
Anaemia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 11
Palpitations (Cardiac disorders) | 3
Hypothyroidism (Endocrine disorders) | 7
Abdominal distention (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 12
Cheilitis (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 13
Dental caries (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 27
Dysphagia (Gastrointestinal disorders) | 4
Haemorrhoids (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 21
Stomatitis (Gastrointestinal disorders) | 29
Vomiting (Gastrointestinal disorders) | 12
Asthenia (General disorders) | 4
Fatigue (General disorders) | 37
Malaise (General disorders) | 7
Oedema peripheral (General disorders) | 14
Pyrexia (General disorders) | 6
Hepatic function abnormal (Hepatobiliary disorders) | 6
Contrast media allergy (Immune system disorders) | 3
Cystitis (Infections and infestations) | 3
Gingivitis (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 14
Paronychia (Infections and infestations) | 5
Pneumonia (Infections and infestations) | 6
Contusion (Injury, poisoning and procedural complications) | 4
Alanine aminotransferase increased (Investigations) | 5
Amylase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 6
Blood bilirubin increased (Investigations) | 5
Electrocardiogram QT prolonged (Investigations) | 4
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 3
Weight decreased (Investigations) | 16
White blood cell count decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 39
Dehydration (Metabolism and nutrition disorders) | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 7
Hyponatraemia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 19
Back pain (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 12
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Dysgeusia (Nervous system disorders) | 5
Headache (Nervous system disorders) | 13
Insomnia (Psychiatric disorders) | 9
Proteinuria (Renal and urinary disorders) | 31
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 10
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 9
Dry skin (Skin and subcutaneous tissue disorders) | 4
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 39
Rash (Skin and subcutaneous tissue disorders) | 10
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 46
Skin infection (Infections and infestations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other